CLINICAL TRIAL: NCT01730469
Title: An Open-Label Study to Determine the Safety and Pharmacokinetics of AT1001 in Subjects With Impaired Renal Function and Healthy Subjects With Normal Renal Function (AT1001-015)
Brief Title: Safety and Pharmacokinetics of AT1001 (Migalastat HCl) in Healthy Subjects and Subjects With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116431
Record Dates: First submitted 2012-11-08; First posted 2012-11-21 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Fabry Disease
Keywords: Pharmacokinetics; GR181413; Safety; AT1001; Migalastat hydrochloride
MeSH Terms: conditions — Fabry Disease | interventions — larazotide acetate; migalastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AT1001 150 mg (Experimental): Each subject will receive a single oral dose of AT1001 150 mg administered orally with 240 mL room temperature water after at least a 4-hour fast
  Interventions: Drug: AT1001 150 mg

INTERVENTIONS:
Drug: AT1001 150 mg — AT1001 150mg is available as a capsule
  Other Names: migalastat HCl; GR181413A

SUMMARY:
This study will assess the safety, tolerability, and pharmacokinetics (PK) study of a single dose of 150 mg AT1001 (migalastat HCl, GR181413A) administered orally to healthy subjects with normal renal function and to subjects with mild, moderate, and severe renal impairment.

DETAILED DESCRIPTION:
This will be an open-label, non-randomized, multiple-center, sequential group, safety, tolerability, and PK study of a single dose of AT1001 (migalastat HCl, GR181413A) administered orally as a 150 mg dose in fasted healthy control male and female subjects with normal renal function compared to mild, moderate, and severe renally-impaired subjects (classified by level of creatinine clearance [CLcr] as determined by the Cockcroft-Gault formula).

Screening will occur from Day -28 to Day -2. Subjects will check-in to the clinic on Day -1 and receive a single oral dose of 150 mg AT1001 on Day 1. Subjects will be discharged from the clinic on Day 2 (if stable as determined by the Investigator) and return for daily visits on Day 3 through Day 6 for a safety assessment and PK sampling. Subjects will undergo a follow-up visit on Day 7 (+1) and an end of study visit on Day 10 (+1).

ELIGIBILITY:
Inclusion Criteria All subjects

* males or females aged 18 to 70 years inclusive (subjects with normal renal function, mild or moderate renal impairment), and 18 to 75 years inclusive (subjects with severe renal impairment)
* body mass index 18.0 to 40.0 kilogram (kg)/square meter (m^2) inclusive
* females who are non-pregnant, non-lactating, or postmenopausal for >=1 year, surgically sterile for >= 90 days, or agree to use approved methods of contraception
* males will be sterile or use approved methods of contraception
* understands and signs informed consent form Healthy subjects with normal renal function
* negative test for selected drugs of abuse (excludes alcohol) at Screening and Check-in
* good health with no clinically significant medical history, physical examination, vital signs, or 12-lead ECG
* clinical laboratory tests within the reference range or not clinically significant
* normal renal function (estimated CLcr >90 mL/min) at Screening Subjects with mild, moderate or severe renal impairment
* negative test for selected drugs of abuse (excludes alcohol) at Screening and Check-in or verification of a prescription for a positive test
* renal impairment (estimated CLcr <90 mL/min)
* evidence of stable renal impairment defined as two separate estimated CLcr values within 25%
* clinical laboratory results consistent with their renal condition or of no clinical significance for the study
* abnormal laboratory values must not be clinically significant. Anemia secondary to renal disease is acceptable if hemoglobin is ≥9 g/dL and no clinically significant symptoms. Liver enzymes and bilirubin must be below twice the upper normal level
* subjects with renal impairment must have stable underlying medical conditions < 90 days before study start
* stable medication regimen(s) (no new drug(s) or changed dosage(s) <30 days before study drug)
* in good general health, allowing for concurrent illnesses associated with chronic kidney disease

Exclusion Criteria:

All subjects:

* history of hypersensitivity or allergies to any drug, unless approved by the Investigator and reviewed by Sponsor/Medical Monitor
* participation in a study with receipt of an investigational drug < 5 half-lives or 30 days (whichever is longer) before Check-in
* use of alcohol, grapefruit, or caffeine-containing foods or beverages < 72 hours before Check-in, unless approved by the Investigator and reviewed by the Sponsor/Medical Monitor
* poor peripheral venous access
* whole blood donation < 56 days before dosing or plasma donation < 14 days before dosing
* receipt of blood products < 2 months before Check-in
* history or presence of any clinically significant abnormal ECG
* history of alcoholism or drug addiction < 1 year before Check-in
* positive test for HIV antibody, HBsAg or anti-HCV
* pregnant or breastfeeding

Healthy subjects with normal renal function:

* use of any tobacco- or nicotine-containing products < 6 months before Check-in
* clinically significant (history of or active) cardiac, hepatic, pulmonary, endocrine, neurological, infectious, gastrointestinal, hematologic, oncologic, or psychiatric disease putting the subject at increased risk or could interfere with study objectives
* screening laboratory values outside normal range and deemed clinically significant by the Investigator
* use of a prescription drug < 14 days of dosing or a non-prescription drug < 7 days before dosing or need of concomitant medication during the study

Subjects with mild, moderate, or severe renal impairment:

* unstable disease (concurrent medical conditions that have changed significantly < 90 days)
* changes in concomitant prescription medications < 30 days before dosing or expected changes during study
* use of new non-prescription medication < 30 days before dosing
* renal transplant
* acute or chronic non-renal condition limiting the subject's ability to complete and/or participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events to assess safety and tolerability | Day 1 to Day 10 (+1)
  Adverse events will be evaluated from Day 1 to the end of study (Day 10 +1).
Clinical laboratory test values to assess safety and tolerability | Day -28 to Day 10 (+1)
  Clinical laboratory evaluations (hematology, clinical chemistry, urinalysis, Hepatitis A and HIV screen) will be evaluated from screening to the end of the study.
Vital signs to assess safety and tolerability | Day -28 to Day 10 (+1)
  Vital signs (oral temperature, respiratory rate, and seated blood pressure) will be performed from screening to the end of the study.
Physician examination to assess safety and tolerability | Day -28 to Day 10 (+1)
  Physical examination (general appearance, skin, thorax/lungs, cardiovascular and abdomen) will be performed from screening to the end of the study.
Measure of ECG to assess safety and tolerability | Day -28 to Day 10 (+1)
  Electrocardiogram (ECG) measures the electrical activity of the heart and the hearts' rhythm. All subjects will undergo ECG testing.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of AT1001 | Day 1 to Day 6
  Blood samples will be collected at predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 15, 24, 48, 72, 96, and 120 hours post-dose and the resultant maximum plasma concentration (Cmax) will be measured in subjects with impaired renal function and normal renal function.
Time to achieve maximum concentration (Tmax) of AT1001 | Day 1 to Day 6
  Blood samples will be collected at predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 15, 24, 48, 72, 96, and 120 hours post-dose and time to maximum concentration (tmax) will be measured in subjects with impaired renal function and normal renal function.
Apparent terminal elimination half life (t1/2 ) of AT1001 | Day 1 to Day 6
  Blood samples will be collected at predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 15, 24, 48, 72, 96, and 120 hours post-dose and and apparent terminal elimination half-life (t1/2) will be measured in subjects with impaired renal function and normal renal function.
Area under the concentration-time curve from time zero to the last measurable concentration (AUC 0-t ) of AT1001 | Day 1 to Day 6
  Blood samples will be collected at predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 15, 24, 48, 72, 96, and 120 hours post-dose and AUC 0-t will be measured in subjects with impaired renal function and normal renal function
Area under the concentration-time curve extrapolated to infinity (AUC 0-inf) of AT1001 | Day 1 to Day 6
  Blood samples will be collected at predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 15, 24, 48, 72, 96, and 120 hours post-dose and AUC 0-inf will be measured in subjects with impaired renal function and normal renal function
Apparent terminal elimination rate constant for AT1001 | Day 1 to Day 6
  Blood samples will be collected at predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 15, 24, 48, 72, 96, and 120 hours post-dose and the apparent terminal elimination rate constant will be measured in subjects with impaired renal function and normal renal function
Oral clearance of AT1001 | Day 1 to Day 6
  Blood samples will be collected at predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 15, 24, 48, 72, 96, and 120 hours post-dose and the oral clearance will be measured in subjects with impaired renal function and normal renal function
Oral volume of distribution of AT1001 | Day 1 to Day 6
  Blood samples will be collected at predose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 15, 24, 48, 72, 96, and 120 hours post-dose and the oral volume of distribution will be measured in subjects with impaired renal function and normal renal function

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (3):
- United States (3):
  - GSK Investigational Site, Costa Mesa, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida

REFERENCES:
- [Derived] Johnson FK, Mudd PN Jr, DiMino T, Vosk J, Sitaraman S, Boudes P, France N, Barlow C. An open-label study to determine the pharmacokinetics and safety of migalastat HCl in subjects with impaired renal function and healthy subjects with normal renal function. Clin Pharmacol Drug Dev. 2015 Jul;4(4):256-61. doi: 10.1002/cpdd.149. Epub 2014 Dec 22. PMID 27136905